CLINICAL TRIAL: NCT03652714
Title: The Effect of Ganglion Sphenopalatine Block (GSP-block) Versus Placebo on Postdural Puncture Headache: a Blinded Randomized Clinical Trial
Brief Title: The Effect of Ganglion Sphenopalatine Block (GSP-block) Versus Placebo on Postdural Puncture Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Mads Seit Jespersen, MD, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSPB-2018
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Postdural Puncture Headache; Sphenopalatine Ganglion Block
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthetic (Experimental)
  Interventions: Procedure: Ganglion sphenopalatine block with local anesthetic
- Isotonic NaCl (Placebo Comparator)
  Interventions: Procedure: Ganglion sphenopalatine block with placebo

INTERVENTIONS:
Procedure: Ganglion sphenopalatine block with local anesthetic — Block performed with bilaterally inserted q-tips with 1:1 mixture of lidocaine 40mg/ml and ropivacaine 5mg/mL.
  Arms: Local anesthetic
Procedure: Ganglion sphenopalatine block with placebo — Block performed with bilaterally inserted q-tips with isotone NaCl
  Arms: Isotonic NaCl

SUMMARY:
The purpose of this study is to evaluate the effect of the ganglion sphenopalatine block (GSP block) on postdural puncture headache.

DETAILED DESCRIPTION:
Adult patients with postdural puncture headache will be enrolled in the study. The patients will be randomised to receive a ganglion sphenopalatine block (GSP-block) with either local anesthetic (lidocaine + ropivacaine) or placebo (isotone NaCl).

Primary outcome is hyperactivity in the sphenopalatine ganglion assessed by pain intensity (0-100mm on a visual analogue scale, VAS) of the postdural headache in standing position 30 minutes after block.

If the patients in the timeframe of 1 hour to 1 week after block does not achieve remission (VAS <30mm while standing) they will be offered a "rescue GSP-block" defined as a new GSP-block with "open-label" local anesthetic and if continued lack of remission at least 1 hour thereafter then an epidural blood patch will be offered.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with postdural puncture headache defined as moderate to severe postural headache (VAS >= 30mm) after lumbar puncture or accidental dural puncture during epidural insertion with an onset within 3 days following the puncture.
* Lack of headache remission within 1 day after dural puncture and after treatment with fluids, caffeine and paracetamol
* Patients who have given their written informed consent for participation in the study after fully understanding the protocol content and limitations.

Exclusion Criteria:

* Patients who cannot cooperate to the study
* Patients who does not understand or speak Danish
* Allergy to the drugs used in the study
* Has taken opioids within 12 hours prior to intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Hyperactivity in the sphenopalatine ganglion assessed by pain intensity (0-100mm on a visual analogue scale, VAS) of the postdural headache in standing position. | 30 minutes after block
  Pain intensity will be measured as worst experienced pain after the patient has been standing for 30 seconds or the worst experienced pain while attempting to stand if the rating has to be interrupted.

SECONDARY OUTCOMES:
Pain rating (0-100mm on a visual analogue scale, VAS) in standing position | 1 hour after block and 1 week after block
  Pain intensity measured as worst experienced pain after the patient has been standing for 30 seconds or the worst experienced pain while attempting to stand if the rating has to be interrupted.
Number of patients with pain rating below 30mm in standing position (0-100mm on a visual analogue scale, VAS) | 30 minutes after block
  Pain intensity measured as worst experienced pain after the patient has been standing for 30 seconds or the worst experienced pain while attempting to stand if the rating has to be interrupted.
Number of patients needing "rescue GSP-block" | During study period until completion of 1 week follow up
Number of patients needing a epidural blood patch | During study period until completion of 1 week follow up
Pain rating (0-100mm on a visual analogue scale, VAS) in supine position | 30 minutes after block, 1 hour after block and 1 week after block

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Rigshospitalet, University of Copenhagen, Copenhagen
  - Bispebjerg and Frederiksberg Hospital, University of Copenhagen, Copenhagen
  - Rigshospitalet Glostrup, University of Copenhagen, Glostrup Municipality
  - Herlev Hospital, University of Copenhagen, Herlev
  - Nordsjællands Hospital Hillerød, Hillerød

REFERENCES:
- [Derived] Jespersen MS, Jaeger P, AEgidius KL, Fabritius ML, Duch P, Rye I, Afshari A, Meyhoff CS. Sphenopalatine ganglion block for the treatment of postdural puncture headache: a randomised, blinded, clinical trial. Br J Anaesth. 2020 Jun;124(6):739-747. doi: 10.1016/j.bja.2020.02.025. Epub 2020 Apr 15. PMID 32303377